CLINICAL TRIAL: NCT06891755
Title: Bronchoscopic RElease of Air Trapped in Hyperinflated Emphysematous Lung - Study 3
Acronym: BREATHE-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Apreo Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0028
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COPD; Emphysema
Keywords: Apreo; COPD; Emphysema; BREATHE System; Hyperinflation; Air-trapping; Apreo BREATHE Airway Scaffold; BREATHE Implant; Airway Scaffold; Apreo Health
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two arm, parallel group, concurrently controlled, open-label, multi-center clinical trial following subjects to 3 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Apreo implants + Optimal Medical Management (Experimental): Treatment group participants will receive optimal medical management and will undergo a single bronchoscopy with bilateral placement of up to 3 implants per lung in appropriately selected targeted airways.
  Interventions: Device: Apreo BREATHE Airway Scaffold
- Optimal Medical Management (Other): Control group participants will receive optimal medical management tailored to patient needs and per standard of care and as outlined in the 2024 GOLD report. This may include smoking cessation, vaccination, long-acting bronchodilator therapy, corticosteroids (when appropriate), and participation in or maintenance of an exercise program or pulmonary rehabilitation program.
  Interventions: Other: Optimal Medical Management (OMM)

INTERVENTIONS:
Device: Apreo BREATHE Airway Scaffold — The experimental treatment involves placement of up to 6 Apreo BREATHE Airway Scaffolds (up to 3 per lung), in a single procedure using bronchoscopy and fluoroscopy. Treatment group subjects will also receive optimal medical management (OMM).
  Arms: Apreo implants + Optimal Medical Management
Other: Optimal Medical Management (OMM) — Subjects will receive optimal medical management tailored to patient needs and per standard of care and as outlined in the 2024 GOLD report. This may include smoking cessation, vaccination, long-acting bronchodilator therapy, corticosteroids (when appropriate), and participation in or maintenance of an exercise program or pulmonary rehabilitation program.
  Arms: Optimal Medical Management

SUMMARY:
The objective of this study is to assess the safety and efficacy of Apreo BREATHE system when used to support native airways and release trapped air in the treatment of adult COPD patients with emphysema suffering from dyspnea due to hyperinflation despite optimal medical treatment. The Apreo BREATHE Airway Scaffold is a permanent implant designed to tent open native airways. The study will include up to 250 participants at up to 25 study centers located in the United States and Europe. Study subjects will be followed for 3 years. The main questions it aims to answer are: Is it safe? Does it work?

DETAILED DESCRIPTION:
Prospective, randomized, two arm, parallel group, concurrently controlled, open-label, multi-center clinical trial following up to 250 participants to 3 years.

Each site will participate in a Roll-In phase prior to participation in the randomized phase of the study. Each site will enroll up to 2 subjects in this phase. Up to 50 subjects may be enrolled into the Roll-In cohort.

Up to 200 subjects with bilateral emphysema will be randomized at up to 25 centers in the United States centers and Europe.

In the Randomized cohort, subjects will be randomized to either a Treatment or Control group in a 2:1 ratio.

* Optimal Medical Management: All subjects (Roll-in and Randomized) will receive optimal medical management tailored to patient needs and per standard of care and as outlined in the 2024 GOLD report. This may include smoking cessation, vaccination, long-acting bronchodilator therapy, corticosteroids (when appropriate), and participation in or maintenance of an exercise program or pulmonary rehabilitation program.
* Treatment group: 133 subjects will receive optimal medical management and Apreo Implant placements. Treatment group subjects will undergo a single bronchoscopy with bilateral placement of up to 3 implants per lung in appropriately selected target airways. Appropriate target segments shall be based on segmental and lobar information (i.e. airway dimensional, emphysematous destruction, volumetric information, hetero/homogeneity) provided in the Quantitative CT (QCT) report for each patient.
* Control group: 67 subjects will receive optimal medical management. Control group subjects will be allowed the opportunity to cross over and receive the BREATHE treatment after their Month 12 visit and within 15 months from their baseline visit.

Subjects will undergo follow-up assessments at Months 1, 3, 6 and 12, and Years 2 and 3 post-procedure (treatment group) or post-randomization (control group). These visits will involve adverse event assessment, questionnaires, pulmonary function testing, and inspiratory/ expiratory CT scans.

Control group subjects electing crossover will then have additional follow-ups at 7- and 30-days post procedure, and 6 months post procedure. Control group subjects not electing crossover will be exited from the study after Month 12.

ELIGIBILITY:
* Inclusion Criteria

  1. Subject is at least 40, but not older than 84, years of age.
  2. Subject has body mass index (BMI) of between 18 and 32, inclusive.
  3. Subject has completed a documented pulmonary rehabilitation program within 12 months prior to Baseline.
  4. Subject has mMRC score ≥ 2.
  5. Subject can walk ≥100 meters in 6 minutes.
  6. Subject has ≥25% emphysema destruction score in each lung as quantified on baseline HRCT scan (low attenuation area less than -950HU) as determined by the CT core lab.
  7. Subject has homogeneous or heterogeneous emphysema, and at least one lung has a 15% difference between upper and lower lobes in emphysema destruction score (-910HU) as determined by the CT core lab.
  8. Subject has bilateral heterogenous emphysema and pre-procedure post-bronchodilator RV ≥ 180% predicted, or one lung with homogenous emphysema and pre-procedure postbronchodilator RV ≥ 200% predicted.
  9. Subject has pre-procedure post-bronchodilator FEV1/ FVC < 0.70.
  10. Subject has a pre-procedure post-bronchodilator FEV1 percent predicted of ≥15% and ≤45%.
  11. Subject has pre-procedure post-bronchodilator RV/TLC ≥ 0.55.
  12. Subject has pre-procedure DLCO ≥ 20%.
  13. Subject has been receiving optimal medical management tailored to subject needs for 2 months prior to enrollment.
  14. Subject has not actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 4 months, and agrees to smoking cessation during the study.
  15. Subject has received preventative vaccinations (or documented clinical intolerance) against potential respiratory infections, including pneumococcus, influenza, RSV (subjects >60 yrs. old) and Covid-19, consistent with local recommendations or policy.
  16. In the opinion of the Primary investigator, subject can undergo bronchoscopy under general anesthesia and is able to adhere to the study follow-up schedule.
  17. Subject has provided written informed consent.
* Exclusion Criteria

  1. Subject has known unresolved lower respiratory tract infection (e.g., pneumonia, mycobacterium avium-intracellulare infection (MAI), fungus, tuberculosis).
  2. Subject has a steroid-dependent condition requiring (e.g. ≥10 mg oral corticosteroid per day).
  3. Subject has bilateral lobar emphysematous destruction scores of >70% percent of voxels with <-950 Hounsfield units on thin slice inspiratory CT, as determined by the CT core lab.
  4. Subject has arterial or capillary blood on room air: PaCO2 > 50 mmHg (8 kPa) or PaO2 ≤ 45 mmHg (6 kPa).
  5. Subject has had ≥2 hospitalization for acute exacerbations of COPD or ≥3 moderate exacerbations/respiratory infections in the year prior to enrollment.
  6. Subject has had previous lung volume reduction surgery, lobectomy, pneumonectomy, segmentectomy, bullectomy, lung transplantation, vapor, glue, or other pulmonary device implant (unless the device has been removed at least 3 months prior to consent).
  7. Subject has known or suspected history of pulmonary arterial hypertension (e.g. PASP > 50mmHg on echocardiogram in absence of confirmation on a right heart catheterization or mPAP > 25mmHg on a right heart catheterization).
  8. Subject has presence of a giant bulla (≥ 30% of hemithorax).
  9. Subject has significant symptom burden due to currently active adult asthma based on GINA criteria and/or chronic bronchitis as their primary diagnosis.
  10. Subject has presence of suspicious radiological abnormalities on HRCT scan such as pulmonary nodule/infiltrate that in judgement of the PI, may require intervention during course of the study.
  11. Subject has clinically significant bronchiectasis (>4 TBS / 45mL mucus production/day, per subject estimate) influencing subject's COPD symptoms.
  12. Subject has unresolved lung cancer.
  13. Subject has a serious medical condition that, in the Primary investigator's opinion, could compromise patient safety or confound the interpretation of the patient's response to therapy (e.g., congestive heart failure, cardiomyopathy (documented LVEF ≤40%), or myocardial infarction in the past year, renal failure, liver disease cerebrovascular accident within the past 6 months, uncontrolled diabetes (HbA1c >8%), uncontrolled hypertension (diastolic BP >110 mmHg or systolic >200 mmHg) or autoimmune disease requiring treatment with immunosuppressant medications or a disease requiring chemotherapy.
  14. Subject is on anticoagulant or antiplatelet therapy for cardiovascular indications and, at the discretion of the Primary investigator, is unable to have anticoagulants withheld for a bronchoscopy procedure per institution's standard of care.
  15. Subject has invasive mechanical ventilator dependency.
  16. Subject is pregnant, lactating, or of childbearing potential and plans to become pregnant during study duration.
  17. Subject has known hypersensitivity to Nitinol (nickel-titanium alloy) or its constituent metals (nickel or titanium).
  18. Subject is significantly immunocompromised, such as organ transplant recipients, those with congenital immune deficiencies, AIDS, or severe rheumatoid arthritis.
  19. Subject has sensitivity or allergy to medications necessary for bronchoscopy under general anesthesia.
  20. Subject is currently participating in another study involving an investigational product that could confound the study results or affect the subject's COPD symptoms.
  21. Subject has within the 2 years prior to consent, had a severe respiratory infection with SARS-CoV-2 (COVID-19) that required ICU support with non-invasive and/or invasive mechanical ventilation.

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) Responder | Month 12
  Defined as a subject who experiences a reduction from baseline in post-bronchodilator FEV1 of ≥12%

SECONDARY OUTCOMES:
Residual Volume (RV) + St George's Respiratory Questionnaire for COPD (SGRQ-C) | Months 3 and 12
  Responder rate
St. George's Respiratory Questionnaire for COPD (SGRQ-C) Responder Rate | Months 3, 6, 12 and Years 2, 3
  SGRQ-C total score
Modified Medical Research Council (mMRC) Responder Rate | Months 3, 6, 12 and Years 2, 3
  mMRC dyspnea score
COPD Assessment Test (CAT) Responder Rate | Months 3, 6, 12 and Years 2, 3
  CAT Score
Forced Expiratory Volume in the first second (FEV1) Responder Rate | Months 3, 6, 12 and Years 2, 3
  FEV1
6-minute walk distance (6MWD) | Months 3, 6, 12 and Years 2, 3
  6MWD
Ratio of residual volume (RV)/ total lung capacity (TLC) Responder Rate | Months 3, 6, 12 and Years 2, 3
  Ratio RV/TLC
Residual Volume (RV) Responder Rate | Months 3, 6, 12 and Years 2, 3
  RV
Forced Vital Capacity (FVC) Responder Rate | Months 3, 6, 12 and Years 2, 3
  FVC

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University
Locations (19):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Health, Gilbert, Arizona
  - University of California at Davis, Sacramento, California
  - Mayo Clinic, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - OSF St Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Clinical Research Associates of Central Pennsylvania, DuBois, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist/Primary Critical Care, Houston, Texas
  - Inova Health Care Services, Falls Church, Virginia
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No